CLINICAL TRIAL: NCT03825640
Title: Project CARE (Community Treatment Adherence at Re-Entry): An Integrated Treatment Adherence Program for Bipolar Disorder at the Time of Prison Release - Open Trial
Brief Title: Project CARE: An Integrated Treatment Adherence Program for Bipolar Disorder at the Time of Prison Release - Open Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1806002090; R34MH117198 (NIH)
Record Dates: First submitted 2019-01-30; First posted 2019-01-31 (Actual); Results first posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2020-02

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Community treatment Adherence at Re-Entry (CARE) (Experimental): CARE will begin within the 2 months before prison release, and will continue for 6 months after re-entry. CARE will be comprised of: a) 3 individual sessions with the CARE counselor; b) 1 optional family/significant other (SO) session; and c) 11 brief (15-20 min) follow-up telephone contacts with prisoners and their SO over the first 6 months post-release.
  The CARE intervention will incorporate motivational strategies from existing interventions (e.g., Acceptance and Commitment Therapy) in order to clarify values and goals to enhance motivation for community treatment engagement and behavior change. CARE will also integrate bipolar disorder psychoeducation and strategies from existing family models of intervention for BD (e.g., McMaster Model of Family Functioning) that are designed to improve family communication, social support, and problem-solving around BD illness management over this vulnerable transition period.
  Interventions: Behavioral: CARE

INTERVENTIONS:
Behavioral: CARE — Hybrid in-person and telephone-based adjunctive intervention for bipolar disorder across the transition from prison to the community.

SUMMARY:
The aim of this program of research is to develop and pilot the CARE (Community treatment Adherence at Re-Entry) program, an adjunctive intervention for incarcerated individuals with bipolar disorder (BD) transitioning from prison to the community.

The purpose of this proposed project is to establish the feasibility, acceptability, and preliminary effects of this newly developed intervention on symptom outcomes.

DETAILED DESCRIPTION:
Bipolar disorder (BD) is a serious, disabling, and highly recurrent illness that is disproportionately represented in the criminal justice system. BD increases risk for several adverse outcomes for prisoners, including mood instability, suicide attempts, substance use relapse, and high rates of repeat incarceration. Despite these serious negative consequences, up to 70% of prisoners with BD do not receive mental health treatment upon prison release. Lack of engagement in ongoing mental health treatment for BD upon community re-entry represents one potent factor that perpetuates risk for adverse outcomes, and consequences of untreated BD (e.g., impulsivity, substance use) may greatly exacerbate difficulties in establishing stable living conditions (e.g., adequate housing, legal employment) at community re-entry. Thus, there is a critical need for interventions to facilitate engagement with treatment for BD during this vulnerable transition.

To that end, the primary aim of this study is to develop and establish the feasibility and acceptability of the Community treatment Adherence at Re-Entry (CARE) program. CARE is an innovative intervention that will combine evidence-based cognitive-behavioral, family, and telephone outreach strategies to promote treatment engagement and improve clinical outcomes for prisoners with BD during the period of community re-entry. CARE will include 3 individual and 1 family session, followed by 11 brief telephone contacts for up to 6 months post-release. Given its moderate intensity, adjunctive nature, use of community mental health counselors, and use of telephone administration for post-release follow-up, CARE has been designed with an eye toward community implementation. Its proposed mechanisms of action (i.e., increasing values-action consistency, enhancing social supports, and linkage to community treatment services) are further well matched to the practical and clinical needs of re-entering individuals.

The aim of this research is to conduct a small open trial (n=12) of the CARE intervention. Assessments will occur at baseline, immediately pre-release, 4 weeks post-release, and 24 weeks post-release (post-treatment). This study will examine the feasibility and acceptability of CARE (e.g., uptake, adherence to, and completion of the CARE intervention, satisfaction with the intervention, understanding of intervention principles) and of this research design. This study will also examine treatment effects (within relevant confidence intervals) on outcomes (e.g., mood symptoms). Change in potential mechanisms (i.e., values-action consistency derived from intervention principles) will be examined.

ELIGIBILITY:
Inclusion Criteria:

* DSM-5 diagnosis of bipolar I, bipolar II, or bipolar disorder not elsewhere classified
* Anticipated prison release within 4-10 weeks
* Expected release to locations anywhere within RI or to locations in other states within a 30 mile radius of Providence
* Aged 18 or older
* Willingness to sign an informed consent document that describes study procedures

Exclusion Criteria:

* Presence of current psychiatric symptoms severe enough to warrant separation from the general prison population
* Cognitive impairment sufficient to prevent successful completion of the baseline interview.
* Inability to understand sufficiently well to understand the consent form or assessment instruments when they are read aloud.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Weinstock, PhD, Principal Investigator — Brown University
Locations (2):
- United States (2):
  - Rhode Island Department of Corrections, Cranston, Rhode Island
  - Brown University, Providence, Rhode Island

RESULTS

PARTICIPANT FLOW:
Groups:
- Community Treatment Adherence at Re-Entry (CARE): CARE will begin within the 2 months before prison release, and will continue for 6 months after re-entry. CARE will be comprised of: a) 3 individual sessions with the CARE counselor; b) 1 optional family/significant other (SO) session; and c) 11 brief (15-20 min) follow-up telephone contacts with prisoners and their SO over the first 6 months post-release.
  The CARE intervention will incorporate motivational strategies from existing interventions (e.g., Acceptance and Commitment Therapy) in order to clarify values and goals to enhance motivation for community treatment engagement and behavior change. CARE will also integrate bipolar disorder psychoeducation and strategies from existing family models of intervention for BD (e.g., McMaster Model of Family Functioning) that are designed to improve family communication, social support, and problem-solving around BD illness management over this vulnerable transition period.
  CARE: Hybrid in-person and telephone-based adjunctive intervention for bipolar disorder across the transition from prison to the community.
- Significant Others (SOs): Significant Others (SOs) are enrolled to support the participant in their study treatment (CARE). SOs only participate in family sessions and brief phone sessions (as described in the CARE arm). SO enrollment is optional.
Period: Overall Study
Arm/Group | Community Treatment Adherence at Re-Entry (CARE) | Significant Others (SOs)
Started | 12 | 6
Completed | 11 | 6
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Community Treatment Adherence at Re-Entry (CARE) | Significant Others (SOs) | Total
Number analyzed (Participants) | 12 | 6 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.08 (11.33) | 48.67 (17.18) | 39.97 (12.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 7 | 2 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 11 | 6 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 8 | 4 | 12
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 12 | 6 | 18

OUTCOME MEASURES:

1. Primary Outcome: Client Satisfaction Questionnaire-8 (CSQ-8)
Description: Intervention feasibility and acceptability. Total Client Satisfaction Questionnaire-8 (CSQ-8) scores range from 8 to 32 with higher scores indicating higher levels of satisfaction.
Time Frame: 24 weeks post-release
Population: Note: 11 of the 12 participants completed the intervention, but one of those individuals was lost to follow-up at the final assessment. Therefore, the total number of participants analyzed is 10. Additionally, Outcome Measure data was not collected for SOs.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Community Treatment Adherence at Re-Entry (CARE)
Number analyzed (Participants) | 10
score on a scale | 27.90 (3.07)

2. Secondary Outcome: Quick Inventory of Depressive Symptomatology - Self-Report (QIDS-SR)
Description: Depressive symptom severity. Total QIDS-SR depressive symptom severity scores range from 0 to 27 with higher scores indicating more severe depressive symptoms.
Time Frame: 24 weeks post-release
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Community Treatment Adherence at Re-Entry (CARE)
Number analyzed (Participants) | 10
score on a scale | 10.90 (5.53)

3. Secondary Outcome: Altman Self-Rating Scale for Mania (ASRM)
Description: Manic symptom severity. Total Altman Self-Rating Scale for Mania (ASRM) manic symptom severity scores range from 0 to 20 with higher scores indicating more severe symptoms of mania.
Time Frame: 24 weeks post-release
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Community Treatment Adherence at Re-Entry (CARE)
Number analyzed (Participants) | 10
score on a scale | 3.30 (4.76)

ADVERSE EVENTS:
Time Frame: The period from baseline to the 24 week follow-up, up to 8 months.
Description: Adverse Event data was only collected from the main study participants. It was not collected from SOs.
Arm/Group | Community Treatment Adherence at Re-Entry (CARE)
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-20): https://cdn.clinicaltrials.gov/large-docs/40/NCT03825640/Prot_SAP_000.pdf